CLINICAL TRIAL: NCT03128099
Title: Physiology-based Virtual Reality Training for Social Skills in Schizophrenia
Brief Title: Virtual Reality Training for Social Skills in Schizophrenia
Acronym: VR-SS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Sohee Park, Professor of Psychology, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: MH106748
Record Dates: First submitted 2017-04-17; First posted 2017-04-25 (Actual); Results first posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Schizophrenia
Keywords: Social Skills; Social attention; Virtual reality; Eye tracking
MeSH Terms: conditions — Schizophrenia; Social Skills

STUDY DESIGN:
Intervention Model Description: Half the participants play the virtual reality video game for one hour per session (low dose).
  The other half play the virtual reality video game for 2 hours per session (high dose).
  Both groups visit the lab 10 times ( twice a week for 5 weeks)
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are assigned to low or high dose randomly. They do not know which condition they are in. The research staff who assess symptoms before and after training do not know which condition the participant is assigned to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose VR social skills training (Experimental): In the low dose condition, participants play the video game for one hour per session. This is a behavioral intervention study. The intervention is playing the social skills virtual reality game to exercise social skills with avatar characters.
  Interventions: Behavioral: Virtual reality social skills training
- High dose Low dose VR social skills training (Experimental): In the high dose condition, participants play the same video game twice per session (it takes them two hours). This is a behavioral intervention study. The intervention is playing the social skills virtual reality game to exercise social skills with avatar characters.
  Interventions: Behavioral: Virtual reality social skills training
- Healthy Control Participants (No Intervention): 23 healthy control participants were recruited and consented to yield baseline comparison data. These participants did not undergo VR training. Only baseline comparison data were collected.

INTERVENTIONS:
Behavioral: Virtual reality social skills training — Participants play a virtual reality video game involving social interactions with various characters ( avatars) at a bus stop, a cafeteria and a grocery store. The games become progressively more complex as the participant improves task performance. Eye tracking patterns are recorded throughout the game to observe the patterns of social attention
  Other Names: physiology based virtual reality social skills training
  Arms: High dose Low dose VR social skills training; Low dose VR social skills training

SUMMARY:
Social impairments are core features of schizophrenia that lead to poor outcome. Social skills and competence improve quality of life and protect against stress-related exacerbation of symptoms, while supporting resilience, interpersonal interactions, and social affiliation. To improve outcome, we must remediate social deficits. Existing psychosocial interventions are moderately effective but the effort-intensive nature (high burden), low adherence, and weak transfer of skills to everyday life present significant hurdles toward recovery. Thus, there is a dire need to develop effective, engaging and low-burden social interventions for people with schizophrenia that will result in better compliance rates and functional outcome.

The investigators will test the effectiveness of a novel adaptive virtual reality (VR) intervention in improving targeted social cognitive function (social attention, as indexed by eye scanning patterns) in individuals with schizophrenia. VR technology offers a flexible alternative to conventional therapies, with several advantages, including a simplified and low-stress social interaction environment with targeted opportunities to simulate, exercise and reinforce basic elements of social skills in a very wide range of realistic scenarios, and to repeat exposure to naturalistic situations from multiple angles.

DETAILED DESCRIPTION:
Social impairments present a major barrier toward good outcome in schizophrenia (SZ). Social skills and social competence protect against stress-related exacerbation of symptoms while supporting interpersonal interactions and social affiliation that help enhance the quality of life. Improving social functions could lead to better outcome and reduce healthcare costs and societal burden. Pharmacotherapy has shown to be inadequate in improving social impairments in schizophrenia, and although existing psychosocial interventions can be moderately effective, the time- and effort-intensive nature (high-burden), low adherence, and weak transfer of skills to real life present significant hurdles. Thus, there is a strong need to develop effective and low-burden social interventions that can be personalized to optimize learning and increase adherence.

Virtual reality (VR) technology offers a very promising alternative to conventional interventions, with several advantages. Controllable complexity of the VR world provides a simplified and low-stress social interaction environment with targeted opportunities to simulate, exercise and reinforce basic elements of social skills and to repeat exposure to naturalistic situations from multiple angles. Simulation of a wide variety of social situations that allows for targeted practice is crucial for learning and transfer of skills. In our proposed VR system, the capacity for personalized social skills training is achieved by automatic and adaptive feedback, based on the affective and attentional states of the participant in real-time, using closed-loop, emotion-sensing VR technology that integrates physiological signals, eye-tracking data and performance data from the participants to rapidly adjust the task parameters. This approach enables realistic, and adaptive interactions in VR games to provide scaffolded social skills exercises in an engaging and enjoyable manner.

The major aim of this proposal is to implement a personalized VR-based social skills training program with high efficacy for individuals with SZ by capitalizing on innovations in adaptive, emotion-sensing technology, designed to increase engagement and learning. This work will be conducted in two phases. The R21 phase will focus on implementing an adaptive social intervention VR game, optimizing the dose and measuring targeted social cognitive outcome. Upon meeting the milestones of the R21 (see 'Approach'), the R33 project will evaluate the feasibility of recruitment, and retention of SZ participants in a pilot randomized controlled trial (RCT) of VR training compared with an active control condition and assess long-term outcome.

The long-term goal of this proposal is to develop and implement a personalized social intervention method for individuals with schizophrenia that is efficacious, low-burden, enjoyable, and with generalizable and enduring benefits. Within the R21 phase, a physiology-based, closed-loop, adaptive VR task will be developed to determine the optimal dose for improving targeted social functions in individuals with SZ. If these goals are met for the R21 phase, a pilot RCT will be conducted in R33 to compare the social, cognitive, neural effects of adaptive social VR versus an active control condition. Furthermore, the physiological and eye tracking data and the outcome data from both R21 and R33 phases will be used to refine and improve this VR protocol and technology. It is hoped that the results of this study will lead to a large scale RCT in the future, and the implementation of a portable, low-cost and widely available intervention that can be personalized for optimal learning. In short, the investigators will implement an efficacious, engaging, low-burden, VR intervention to ameliorate social impairments of SZ and improve functional outcome.

ELIGIBILITY:
Inclusion and Exclusion Criteria:

Individuals with Schizophrenia:

* DSM-5 Axis 1 Diagnosis of schizophrenia
* No DSM 5 Axis 1 diagnosis other than schizophrenia
* No diagnosed organic brain disease, brain lesions, history of head traumas, neurological disorders or other conditions that involve the degeneration of the central nervous system (e.g. multiple sclerosis)
* No substance/alcohol abuse/dependence during the past 1 year
* No tardive dyskinesia
* WASI IQ> 90
* Currently taking antipsychotic medication
* No change in current psychotropic medications or housing within the past 30 days. Those patients whose medication or housing situation has changed within a month, we will wait list them until their situation stabilizes.

Inclusion and exclusion criteria for the healthy control group:

* No DSM-5 Axis 1 diagnosis of psychotic disorders in themselves or their families (e.g. schizophrenia, bipolar disorder).
* No antipsychotic medications
* No diagnosed organic brain disease, brain lesions, history of head traumas, neurological disorders or other conditions that involve the degeneration of the central nervous system (e.g. multiple sclerosis)
* No substance/alcohol abuse/dependence during the past 1 year
* WAIS IQ > 90.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sohee Park, PhD, Principal Investigator — Vanderbilt University; Nilanjan Sarkar, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Adery LH, Ichinose M, Torregrossa LJ, Wade J, Nichols H, Bekele E, Bian D, Gizdic A, Granholm E, Sarkar N, Park S. The acceptability and feasibility of a novel virtual reality based social skills training game for schizophrenia: Preliminary findings. Psychiatry Res. 2018 Dec;270:496-502. doi: 10.1016/j.psychres.2018.10.014. Epub 2018 Oct 9. PMID 30326433
- [Result] Torregrossa LJ, Bian D, Wade J, Adery LH, Ichinose M, Nichols H, Bekele E, Sarkar N, Park S. Decoupling of spontaneous facial mimicry from emotion recognition in schizophrenia. Psychiatry Res. 2019 May;275:169-176. doi: 10.1016/j.psychres.2019.03.035. Epub 2019 Mar 20. PMID 30921747
- [Result] Wade J, Nichols HS, Ichinose M, Bian D, Bekele E, Snodgress M, Amat AZ, Granholm E, Park S, Sarkar N. Extraction of Emotional Information via Visual Scanning Patterns: A Feasibility Study of Participants with Schizophrenia and Neurotypical Individuals. ACM Trans Access Comput. 2018 Nov;11(4):23. doi: 10.1145/3282434. PMID 30627303
- [Derived] Roberts MT, Lloyd J, Valimaki M, Ho GW, Freemantle M, Bekefi AZ. Video games for people with schizophrenia. Cochrane Database Syst Rev. 2021 Feb 4;2(2):CD012844. doi: 10.1002/14651858.CD012844.pub2. PMID 33539561

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose VR Social Skills Training: In the low dose condition, participants play the video game for one hour per session. This is a behavioral intervention study. The intervention is playing the social skills virtual reality game to exercise social skills with avatar characters.
  Virtual reality social skills training: Participants play a virtual reality video game involving social interactions with various characters ( avatars) at a bus stop, a cafeteria and a grocery store. The games become progressively more complex as the participant improves task performance. Eye tracking patterns are recorded throughout the game to observe the patterns of social attention. Social attention was indexed by a measure called Social Engagement latency (SEL).
- High Dose VR Social Skills Training: In the high dose condition, participants play the same video game twice per session (it takes them two hours). This is a behavioral intervention study. The intervention is playing the social skills virtual reality game to exercise social skills with avatar characters.
  Virtual reality social skills training: Participants play a virtual reality video game involving social interactions with various characters ( avatars) at a bus stop, a cafeteria and a grocery store. The games become progressively more complex as the participant improves task performance. Eye tracking patterns are recorded throughout the game to observe the patterns of social attention. Social attention was indexed by a measure called Social Engagement latency (SEL).
- Healthy Control Participants: Control participants were recruited to obtain normative data
Period: Overall Study
Arm/Group | Low Dose VR Social Skills Training | High Dose VR Social Skills Training | Healthy Control Participants
Started | 21 | 4 | 22
Hour 1 (Low Dose) Started | 21 | 4 | 22
Hour 1 (Low Dose) Completed | 19 | 4 | 21
Hour 2 (High Dose)Started | 0 (Hour 2 of training not available to these participants) | 4 | 0 (Hour 2 of training not available to these participants)
Hour 2 (High Dose) Completed | 0 | 0 | 0
Completed | 19 | 0 (hour 2 training was completed by 0 participants) | 21
Not Completed | 2 | 4 | 1
Not completed — High dose task was too long | 0 | 4 | 0
Not completed — Participant got a full time job. | 1 | 0 | 0
Not completed — Became homeless and lost contact | 1 | 0 | 0
Not completed — Did not complete all the assessments | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- High Dose VR Social Skills Training: In the high dose condition, participants play the same video game twice per session (it takes them two hours). This is a behavioral intervention study. The intervention is playing the social skills virtual reality game to exercise social skills with avatar characters.
  Virtual reality social skills training: Participants play a virtual reality video game involving social interactions with various characters ( avatars) at a bus stop, a cafeteria and a grocery store. The games become progressively more complex as the participant improves task performance. Eye tracking patterns are recorded throughout the game to observe the patterns of social attention
- Healthy Control Participants: Control participants were recruited to provide normative data
- Total: Total of all reporting groups
Arm/Group | Low Dose VR Social Skills Training | High Dose VR Social Skills Training | Healthy Control Participants | Total
Number analyzed (Participants) | 21 | 4 | 22 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.78 (7.42) | 47.52 (10.08) | 45.65 (8.17) | 47.2 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 0 | 12 | 22
  Male | 11 | 4 | 10 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 1 | 0 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 13 | 4 | 5 | 22
  White | 6 | 0 | 14 | 20
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 21 | 4 | 22 | 47
Baseline Social Attention [Mean (Standard Deviation); unit: milliseconds] — Social attention is indexed by Social Engagement Latency (SEL). SEL is defined as the time taken to select an avatar by fixating eye gaze at the chosen avatar's face to initiate a new social 'mission'. SEL is measured in milliseconds. This is an ecologically valid index that corresponds to one's readiness to initiate a social interaction. Population: No participants completed the High dose VR social skills training. The control group did not receive any VR training
  milliseconds
    number analyzed (Participants) | 21 | 0 | 0 | 21
    (all) | 32824 (11932) |  |  | 32824 (11932)

OUTCOME MEASURES:

1. Primary Outcome: Social Attention: Social Engagement Latency (SEL)
Description: Social Engagement Latency (SEL), defined as the time taken to select an avatar by fixating eye gaze at the chosen avatar's face to initiate a new social 'mission'. This is an ecologically valid index that corresponds to one's readiness to initiate a social interaction.
  To start a social 'mission', the participant must choose an avatar by fixating on a semi-transparent green patch that covers the avatar's face. When the participant fixates on the avatar's face, the green patch disappears to reveal the avatar's face, which starts the social mission game.
  The time takes to remove the green patch to reveal the avatar's face is the SEL, our primary social attention target and a useful index of pro-social attention engagement.
Time Frame: 5 weeks
Population: NB: We did not run high dose condition due to the feasibility problem. Control participants do not undergo training. Therefore only the results of the low dose condition are reported
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Low Dose VR Social Skills Training
Number analyzed (Participants) | 18
msec | 21618 (4134)

ADVERSE EVENTS:
Time Frame: The training took 5 weeks but the pre-training baseline data collection and post-training assessment were conducted before and after these 5-week training periods. Therefore potential adverse events were monitored for each participant for between 7 weeks and 10 weeks. There were no adverse events.
Groups:
- Low Dose VR Social Skills Training: In the low dose condition, participants play the video game for 1 hour per session. This is a behavioral intervention study. The intervention is playing the social skills VR game to exercise social skills with avatar characters.
  VR social skills training: Participants play a VR video game involving social interactions with various characters (avatars) at a bus stop, a cafeteria and a store. The games become progressively more complex as the task performance improves. Eye tracking patterns are recorded throughout the game to observe the patterns of social attention
- High Dose VR Social Skills Training: In the high dose condition, participants play the same video game twice per session (2 hours). This is a behavioral intervention study. The intervention is playing the social skills VR game to exercise social skills with avatar characters.
  VR social skills training: Participants play a VR video game involving social interactions with various characters (avatars) at a bus stop, a cafeteria and a store. The games become progressively more complex as the participant improves task performance. Eye tracking patterns are recorded throughout the game to observe the patterns of social attention.
  Please note that because of the burdensome nature of playing this video game for 2 hours, no participant completed this condition. 4 started and completed 1 hour per session ( equivalent to the low dose condition) but they did not play 2 hours per session.
- Healthy Controls: Control participants did not undergo training (no intervention). They were only tested to establish normative baseline test scores.
Arm/Group | Low Dose VR Social Skills Training | High Dose VR Social Skills Training | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/4 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/4 | 0/22
Other Adverse Events (participants affected / at risk) | 0/21 | 0/4 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/99/NCT03128099/Prot_SAP_000.pdf